CLINICAL TRIAL: NCT05986812
Title: Feasibility of Shear Wave Elastography in Assessment of Renal Stiffness in Chronic Kidney Diseased Patients
Brief Title: SWE in Assessment of CKD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina AbdAllah Noshy AbdAllah, Dina AbdAllah, Assiut University
Other Study IDs: Renal Elastography
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Elastography ,CKD Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal subjects
- Diseased subjects

SUMMARY:
Elastography is a developing technique to assess tissue elasticity. It is software that can be integrated to the ultrasonography machines. Shear wave Elastography (SWE) is an Elastography technique that does not require external pressure on the tissue and supplies quantitative data. It uses real-time short-duration acoustic push pulse to generate shear waves that propagate perpendicular to the main ultrasound beam. When the waves hit the targeted tissue, the tissue is "pushed" in the direction of propagation, causing it to temporarily deform or displace. The ultrasound scanner can monitor the tissue displacement, measuring the time-to-peak displacement and the recovery time. Shear wave velocity increases in diseased tissues, which can be significantly stiffer than normal ones. The parameters are expressed in pressure units of kilopascals (kPa) and velocity (m s-1). SWE have been used to study breast, thyroid, prostate and liver diseases. However, the application of SWE in assessment of renal fibrosis in CKD patients is still unclear.

ELIGIBILITY:
Inclusion Criteria:

* The patients are those older than 18 years diagnosed with CKD based on the KDIGO (Kidney Disease Improving Global Outcomes) definition i.e. eGFR less than 60 mL/min and/or the presence of markers of kidney damage (pathological albuminuria of at least 30 mg per 24 hours or proteinuria, hematuria, casts) persisting for more than 3 months.

Exclusion Criteria:

* Patients whose BMI >35kg/m 2 Any condition that precludes visualization of the kidney by ultrasound or transmission of shear waves as pregnancy or marked ascites patients with surgical kidney problems like hydro or pyonephrosis patients unwilling to complete the study. Patients with a history of renal replacement therapy (hemodialysis, peritoneal dialysis) , renal transplant, or acute kidney injury within the last 3 months Patients with cystic kidney disease Patients with renal masses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD patients which ages from 18 to 75 years old
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-10-25 (Estimated); Primary Completion 2024-10-25 (Estimated); Study Completion 2025-10-24 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study is the difference in renal SWE values between normal subjects and CKD patients . | From 2 to 3 years